CLINICAL TRIAL: NCT04284423
Title: Study of Synovial Lactate Level as Marker of Septic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/00501
Record Dates: First submitted 2019-12-30; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Joint fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: joint fluid lactate — Analysis of lactate level in joint fluid to determine presence of septic joint

SUMMARY:
Lactate levels are rapidly available and may potentially aid in diagnosing septic arthritis in a native joint. This study will determine the utility of synovial lactate in discriminating septic from aseptic arthritis.

DETAILED DESCRIPTION:
A painful, swollen joint can be caused by variety of conditions. Distinguishing bacterial arthritis and other causes of arthritis is essential to reducing significant morbidity and mortality. In most cases, septic arthritis is monoarticular and occurs most commonly in large peripheral joints, such as the knee.

Current recommended diagnostic tools include clinical suspicion after examination followed by testing of synovial fluid from the affected joint. The gold standard is often gram stain or synovial fluid culture. The early markers such as synovial WBC, polymorphonuclear white blood cells are not accurate in predicting the diagnosis of septic arthritis. This leads to diagnostic dilemmas, inappropriate admissions, and unnecessary costs pending the results of synovial fluid cultures.

The current emergency department protocol for the diagnosis of septic arthritis states that if none of the following criteria is met, it is unlikely to be septic arthritis:

1. synovial fluid white cell count more than 50 000/uL; or
2. synovial fluid neutrophil more than 75%; or
3. positive gram stain.

However, it has been noted that septic arthritis can have white cell counts lower than 50 000/uL which means that the current protocol cannot safely rule out septic arthritis. A neutrophil percentage of at least 90% has a reported specificity ranging from 68 to 83% while our current protocol uses a cut off of 75% which has a low specificity resulting in many unnecessary admissions. A high neutrophil percentage is also seen in inflammatory joint conditions, and therefore may not be adequate to distinguish infective from non-infective joint pain. A recent review of existing studies in 2011 stated "Future ED-based diagnostic trials are needed to evaluate the role of clinical gestalt and the efficacy of nontraditional synovial markers such as lactate".

The most recent pertinent study was published in Acta Orthopædica Belgica 2014. This was a small retrospective study comparing septic arthritis to aseptic arthritis in samples taken from the emergency department between 2006 and 2013. In the final analysis, lactate was identified as the most accurate early marker in predicting a positive synovial fluid culture. The reported sensitivity was 74.5% with a specificity of 87.2%. This study is limited by its retrospective nature, small sample sizes, and lack of information regarding the prevalence of disease in the local population.

A metanalysis in the Journal of the American Medical Association 2007 cited two studies that reported a prevalence of septic joint in the study population of 8% and 27%. The prevalence of septic joint in our local population is unknown. This study will reveal the incidence of septic joints in the emergency department population.

Review of data from the Khoo Teck Puat Hospital electronic medical records from six months in 2018 reveal 91 synovial joint samples tested for gram stain, culture, or cell count. The investigators expect it will take one year to obtain 200 samples.

ELIGIBILITY:
Inclusion criteria:

* Age 21 and older
* Suspected infected joint

Exclusion criteria:

* Age under 21
* Prosthetic joint affected
* Overlying cellulitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 21 years or older with tender swollen joints undergoing arthrocentesis will be enrolled in the study. Exclusion criteria will be overlying cellulitis, affected prosthetic joints and age under 21.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-08 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Lactate level of synovial fluid | The duration of study is one year.
  Lactate levels of joint fluid of suspected infected knee joint. The gold standard for infected joint will be performance of washout procedure or positive gram stain or culture.

CONTACTS AND LOCATIONS:
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margaretten ME, Kohlwes J, Moore D, Bent S. Does this adult patient have septic arthritis? JAMA. 2007 Apr 4;297(13):1478-88. doi: 10.1001/jama.297.13.1478. PMID 17405973
- [Background] Lenski M, Scherer MA. The significance of interleukin-6 and lactate in the synovial fluid for diagnosing native septic arthritis. Acta Orthop Belg. 2014 Mar;80(1):18-25. PMID 24873080
- [Background] Carpenter CR, Schuur JD, Everett WW, Pines JM. Evidence-based diagnostics: adult septic arthritis. Acad Emerg Med. 2011 Aug;18(8):781-96. doi: 10.1111/j.1553-2712.2011.01121.x. PMID 21843213